CLINICAL TRIAL: NCT06701175
Title: Anterolateral Geniculate Nerve Block and Portal Anesthesia in Knee Arthroscopy for Pain Control: A Randomized Control Trial
Brief Title: Knee Arthroscopy for Pain Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Aaron Casp, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013299; UAB (Other: UAB)
Record Dates: First submitted 2024-11-11; First posted 2024-11-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthroscopy
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Patients indicated for knee arthroscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention (No Intervention): Patients will receive no intervention
- Nerve Block (Active Comparator): Patients in the anterolateral geniculate nerve block group will receive 20 cc of 0.25% bupivacaine with epinephrine distributed evenly between two injection sites by an 18G or 21G long needle. After completion of knee arthroscopy, the first injection is targeted at 2 fingerbreadths superior to the superolateral aspect of the patella. The needle is inserted down to the femur, pulled back slightly, and the surrounding area is infiltrated with 10 cc of anesthetic. The second injection is targeted approximately 2 to 3 fingerbreadths laterally to the first injection and 2 to 3 fingerbreadths proximal to the lateral epicondyle in line with the lateral femur. Once again, the needle is inserted down until bone is encountered and then slightly retracted 1 to 2 mm before infiltration with the remaining 10 cc of anesthetic.
  Interventions: Procedure: Nerve Block
- Portal Anesthesia (Active Comparator): Patients in the portal anesthesia group will also receive 20 cc of 0.25% bupivacaine with epinephrine distributed evenly between portal sites. After completion of knee arthroscopy, portal tracts are closed and the knee is ensured to be evacuated of residual fluid. An 18G or 21G long needle is then used to infiltrate each portal tract where the anesthetic will be delivered.
  Interventions: Procedure: Portal Anesthesia

INTERVENTIONS:
Procedure: Nerve Block — anterolateral geniculate nerve block
  Arms: Nerve Block
Procedure: Portal Anesthesia — portal anesthesia
  Arms: Portal Anesthesia

SUMMARY:
This study aims to determine the effectiveness of an anterolateral genicular nerve block and portal anesthesia in controlling pain in the perioperative period after knee arthroscopy. Opioid consumption, the use of non-opioid medications, complication rate, and sleep quality will also be measured.

DETAILED DESCRIPTION:
Orthopaedic surgeries are some of the most painful operations to recover from, especially when involving cruciate ligaments. Because of this, orthopaedic surgeons have worked to optimize postoperative pain management that provides the best relief. Opioids traditionally were the primary medication for pain control during the perioperative period, however, with the current opioid epidemic and opioids being the leading cause of accidental deaths in the United States, physicians have transitioned to multimodal pain control which has shown to provide better pain control. In cases involving knee arthroscopy, pain management options include variations of nerve blocks, medications, surgical techniques, and postoperative activity.

An anterolateral genicular nerve block has been proposed that focuses on decreasing postoperative pain in the lateral aspect of the knee by targeting the lateral retinacular nerve, the nerve to the vastus lateralis, and the articular branch of the nerve to the vastus intermedius. Adductor canal blocks and intraarticular injections are known methods of providing postoperative pain control, but due to their risks, they may be inappropriate for knee arthroscopy. An anterolateral geniculate nerve block targets sensory, terminal nerve fibers outside the joint capsule, theoretically avoiding the risks of large nerve irritation and chondrotoxicity. Postoperative portal injections are another form of analgesia provided after knee arthroscopy and have been demonstrated to be equally effective in controlling pain as intraarticular injections one hour postoperatively. Otherwise, portal injections in knee arthroscopy have not been extensively studied in the literature.

Patients will be sent home after surgery with a survey to be completed at 2, 4, 6, 12, 24, and 48 hours and 1 week. The survey will inquire about the period from the prior survey to the current survey and will evaluate pain via Visual Analog Score, opioid consumption, non-opioid medication use, sleep, and intervention complications. Patients will be called at 12 and 48 hours and 1 week as reminders to complete the survey.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patients with indications for knee arthroscopy

Exclusion Criteria:

* include patients with previous knee surgery on the operative side
* opioid use within six weeks before surgery that is deemed to be chronic or excessive
* gabapentin use within six weeks before surgery
* diagnosis of chronic pain, fibromyalgia, or other somatosensory disorder(s)
* history of radicular pain or neuropathy in the operative limb
* patients with cancer

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Management | 2, 4, 6, 12, 24, and 48 hours and 1 week post-op
  Collected variables will include average and worst pain (0-10 scale, higher values representing increased pain), dose frequency of prescribed opioid analgesics, consumption of prescribed nonopioid analgesics, the longest period of uninterrupted sleep (in hours; only obtained at 12 and 24 hours and 1 week), and the subjective quality of sleep (0-10 scale, higher values representing better sleep), and overall satisfaction with pain control (five-point Likert scale, higher values representing increased satisfaction). A Visual Analog Score will be used in the evaluation of pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Townshend D, Emmerson K, Jones S, Partington P, Muller S. Intra-articular injection versus portal infiltration of 0.5% bupivacaine following arthroscopy of the knee: a prospective, randomised double-blinded trial. J Bone Joint Surg Br. 2009 May;91(5):601-3. doi: 10.1302/0301-620X.91B5.21932. PMID 19407292
- [Background] Ghodki PS, Shalu PS, Sardesai SP. Ultrasound-guided adductor canal block versus femoral nerve block for arthroscopic anterior cruciate ligament repair under general anesthesia. J Anaesthesiol Clin Pharmacol. 2018 Apr-Jun;34(2):242-246. doi: 10.4103/joacp.JOACP_172_17. PMID 30104837
- [Background] Howell R, Hill B, Hoffman C, Treacy E, Mulcahey MK. Peripheral Nerve Blocks for Surgery About the Knee. JBJS Rev. 2016 Dec 6;4(12):e1. doi: 10.2106/JBJS.RVW.16.00003. PMID 28060787
- [Background] Tyler TF, McHugh MP, Gleim GW, Nicholas SJ. The effect of immediate weightbearing after anterior cruciate ligament reconstruction. Clin Orthop Relat Res. 1998 Dec;(357):141-8. doi: 10.1097/00003086-199812000-00019. PMID 9917711
- [Background] Chunduri A, Aggarwal AK. Multimodal Pain Management in Orthopedic Surgery. J Clin Med. 2022 Oct 28;11(21):6386. doi: 10.3390/jcm11216386. PMID 36362617
- [Background] Paul RW, Szukics PF, Brutico J, Tjoumakaris FP, Freedman KB. Postoperative Multimodal Pain Management and Opioid Consumption in Arthroscopy Clinical Trials: A Systematic Review. Arthrosc Sports Med Rehabil. 2021 Dec 17;4(2):e721-e746. doi: 10.1016/j.asmr.2021.09.011. eCollection 2022 Apr. PMID 35494281
- [Background] Meissner W, Mescha S, Rothaug J, Zwacka S, Goettermann A, Ulrich K, Schleppers A. Quality improvement in postoperative pain management: results from the QUIPS project. Dtsch Arztebl Int. 2008 Dec;105(50):865-70. doi: 10.3238/arztebl.2008.0865. Epub 2008 Dec 12. PMID 19561807